CLINICAL TRIAL: NCT01564797
Title: Partnership for a Hispanic Diabetes Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IR6194
Record Dates: First submitted 2012-03-23; First posted 2012-03-28 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes; Pre-diabetes
Keywords: Diabetes; haemoglobin A1C; Hispanic; Behavioural Intervention
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education Intervention (Active Comparator): A series of 5 home-based lay health educator-led education sessions (Home Health Parties (HHP)), to educate a Hispanic population about diabetes, management of diabetes, and diet and exercise
  Interventions: Behavioral: Home Health Party
- Control Arm (No Intervention): A delayed intervention where the intervention was delivered after the hA1c level was measured for the second time (3 months after the baseline measurement)

INTERVENTIONS:
Behavioral: Home Health Party — An education-based lay health educator-led intervention designed to educate Hispanic participants with elevated HA1c levels about diabetes, treatment of diabetes, and diet and lifestyle changes.
  Arms: Education Intervention

SUMMARY:
The aims of the study are to investigate

1. the effects of an intervention vs. control on levels of glycosylated haemoglobin (haemoglobin A1c) in Hispanic participants, older than 18 years, who have elevated hA1c at baseline (>6.0%). Glycosylated haemoglobin provides an indication of blood sugar levels over the past 3 months. Elevated hA1c levels are seen in diabetics and pre-diabetics.
2. the effects of the intervention vs control on consumption of fresh fruit and vegetables
3. the effects of the intervention vs control on levels of physical activity

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older
* Haemogloblin A1c ≥ 6.5%
* Hispanic Ethnicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2008-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Effect of the intervention on serum levels of hA1c in diabetics and pre-diabetic participants | Baseline, 3 months
  Test the efficacy of an intervention to educate diabetics and pre-diabetics about the management of diabetes as assessed by decreases in hemoglobin A1c;
Effect of the intervention on consumption of fresh fruit and vegetables in diabetics and pre-diabetic participants | Baseline, 3 months
  Test the efficacy of an intervention to increase the consumption of healthy diets as assessed by increases in fruit and vegetable consumption
Effect of the intervention on physical activity levels in diabetics and pre-diabetic participants | Baseline, 3 months
  Test the efficacy of an intervention to increase physical activity as assessed by increases in the times per week engaged in strenuous or moderate activity.

SECONDARY OUTCOMES:
Effect of the intervention on changes in knowledge and attitudes about diabetes | Baseline, 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Beti Thompson, PhD, Principal Investigator — Fred Hutchinson Cancer Center

REFERENCES:
- [Derived] Duggan C, Carosso E, Mariscal N, Islas I, Ibarra G, Holte S, Copeland W, Linde S, Thompson B. Diabetes prevention in Hispanics: report from a randomized controlled trial. Prev Chronic Dis. 2014 Feb 27;11:E28. doi: 10.5888/pcd11.130119. PMID 24576395